CLINICAL TRIAL: NCT06007859
Title: Influence of Section Orientation of Ultrasound Shear Wave Elastography on the Measurement of Thyroid Nodules Stiffness
Brief Title: Patients Who Underwent Thyroid Ultrasonography at Our Institution Were Selected for Shear Wave Elastography of Thyroid Nodules, and the Maximum and Mean Values of the Modulus of Elasticity of the Nodules in Transverse and Longitudinal Sections Were Analyzed.
Acronym: SWE
Status: Completed | Type: Observational
Sponsor: Ma Zhe (Other)
Responsible Party: Sponsor-Investigator, Ma Zhe, Director of Ultrasound, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(024)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Thyroid Nodules
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- section orientation of ultrasound shear wave elastography
  Interventions: Other: section orientation

INTERVENTIONS:
Other: section orientation — The patient was placed in a decubitus supine head back extension position to fully expose the cervical thyroid examination site. The instrument was adjusted appropriately to achieve optimal imaging quality, the suspicious nodule was located in conventional ultrasound mode, the SWE option in VT mode was selected, and the patient was instructed to hold his/her breath to minimize the effect of respiration, and elastograms of the nodule in transverse and longitudinal sections were obtained.

SUMMARY:
The objective of this observational study was to evaluate the effect of transverse and longitudinal sections on the measurement of thyroid nodule stiffness by shear wave elastography. The main questions it aims to answer are: (i) to compare the diagnostic efficacy of different section orientations of shear wave elastography for the diagnosis of benign and malignant thyroid nodules; (ii) to analyze the correlation between the two orientations of transverse and longitudinal sections of shear wave elastography; and (iii) to compare the reliability and consistency of the two orientations of transverse and longitudinal sections of shear wave elastography for the diagnosis of thyroid nodules. Participants will undergo routine ultrasound examination of the thyroid gland and shear wave elastography, and the measured modulus of elasticity of the nodules in both transverse and longitudinal sections will be recorded.

ELIGIBILITY:
Inclusion Criteria:

All patients underwent preoperative shear-wave elastography ultrasonography; thyroid nodules ranged from 3 to 20 mm in size; all nodules underwent puncture biopsy or surgery to obtain pathologic results.

Exclusion Criteria:

Unavailability of pathology results for various reasons; poor quality of ultrasound images; missing data.

Ages: 22 Years to 68 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid nodules attending the First Affiliated Hospital of Shandong First Medical University were selected.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
elastic modulus values | The elastic modulus values of different sections were recorded immediately after the patients underwent routine ultrasound and shear wave elastography and the recorded results were saved.
  the maximum value of elastic modulus (Emax) and the average value of elastic modulus (Emean) of benign and malignant nodules in both longitudinal and transverse sections

CONTACTS AND LOCATIONS:
Locations (1):
- QianfoshanH, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Lack of resources or infrastructure: Sharing IPDs requires resources and infrastructure to ensure data security, manage access requests and provide necessary documentation. Currently these resources are not well developed, so it may be difficult to share IPDs.